CLINICAL TRIAL: NCT05407038
Title: Remote Monitoring With Health-Coaching for Lifestyle Changes in Patients With Lung Cancer Related Fatigue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped early due to enrollment challenges.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-013228; NCI-2022-02155 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-013228 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-06-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (remote monitoring with health coaching) (Experimental): Patients undergo routine exercise using a remote monitoring system (Garmin Vívofit activity monitor, Nonin 3150 WristOx2 pulse oximeter, and an Android tablet) over 30 minutes at least 6 days per week and complete daily questionnaires over 20 minutes for 12 weeks. Patients also receive health coaching telephone calls over 5-20 minutes once a week for 12 weeks. At the end of the 12 weeks, patients complete an audio taped telephone interview.
  Interventions: Other: Exercise Counseling; Other: Exercise Intervention; Other: Internet-Based Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Exercise Counseling — Receive call from health coach
Other: Exercise Intervention — Undergo routine exercise
Other: Internet-Based Intervention — Receive Android tablet
Other: Interview — Complete a qualitative interview
Other: Medical Device Usage and Evaluation — Wear Garmin Vivofit and Nonin 3150 WristOx2 pulse oximeter
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial investigates the effectiveness of a remote monitoring program for lifestyle changes in patients with lung cancer related fatigue (CRF). Fatigue is a common symptom of lung cancer and a side-effect of cancer treatments. CRF has a negative impact on patients' quality of life, daily activities, employment, social relationships and mood. Health coaches enable patients to develop and achieve self-determined wellness goals and assist patients to use their insight, personal strengths, goal setting, action steps, and accountability toward achieving healthy lifestyle changes. Remote monitoring with health-coaching may help relieve lung cancer related fatigue and increase the quality of life in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effect of the remote-monitoring program on patient reported fatigue by administering the Brief Fatigue Inventory (BFI), Functional Assessment of Cancer Therapy Fatigue (FACT-F), Functional Assessment of Cancer Therapy- Lung (FACT-L) and the Modified Fatigue Impact Scale (MFIS).

OUTLINE:

Patients undergo routine exercise using a remote monitoring system (Garmin Vívofit activity monitor, Nonin 3150 WristOx2 pulse oximeter, and an Android tablet) over 30 minutes at least 6 days per week and complete daily questionnaires over 20 minutes for 12 weeks. Patients also receive health coaching telephone calls over 5-20 minutes once a week for 12 weeks. At the end of the 12 weeks, patients complete an audio taped telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced lung non-small cell carcinoma (NSCLC) being treated with any line of non-curative intent, systemic treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 (asymptomatic) to 2.
* The ability to read and respond to questions in English or Spanish
* Receiving primary cancer care at Mayo Clinic, Rochester or Mayo Clinic Health System (MCHS).
* Age > 18 years.
* Life expectancy at least 6 months.
* Moderate or higher fatigue (>= 4) on a scale of 0-10 based on fatigue rating to question: Rate your average fatigue over the last week, where 0 is no fatigue and 10 is extreme fatigue.

Exclusion Criteria:

* They have cognitive or psychiatric conditions as determined by the treating oncologist to prohibit study consent or participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Fatigue | Baseline to 3 months
  The BFI is a nine item questionnaire with a 10 point numeric scale measuring fatigue level and it's interference with daily life. The higher the score the more fatigue.

SECONDARY OUTCOMES:
Quality of life fatigue assessement | Baseline to 3 months
  The functional assessment is a 50 item questionnaire that measures self-reported fatigue and its impact on daily living using a Likert scale from Not at all (0) to Very Much (4).The higher the score the more symptoms interfere with daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P. Benzo, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials